CLINICAL TRIAL: NCT02146911
Title: Evaluating the Real-world Effectiveness of Varenicline and Bupropion for Long-term Smoking Cessation
Brief Title: The MATCH (Medication Aids for Tobacco Cessation and Health) Study
Acronym: MATCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Global Research Awards for Nicotine Dependence (GRAND) (Unknown)
Responsible Party: Principal Investigator, Laurie Zawertailo, Independent Scientist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200/2012
Record Dates: First submitted 2014-05-20; First posted 2014-05-26 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-01

CONDITIONS: Tobacco Use Disorder; Nicotine Dependence
Keywords: Smoking Cessation Medication; Smoking Treatment; Tobacco Treatment; Quitting Smoking; Bupropion; Varenicline; Efficacy; Pharmacogenetics of Smoking Treatment; Genetics analysis; Smoking Personality; Dependence; Addiction; Cigarettes; Primary Care Physicians; Biochemical Confirmation
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation; Behavior, Addictive | interventions — Bupropion; Varenicline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bupropion (Experimental): Bupropion hydrochloride SR, Sandoz Canada, Boucherville, Quebec. Dispense for 12 weeks. One tablet (150mg) once daily for first three days, then twice daily for the remainder of 12 weeks.
  Interventions: Drug: Bupropion; Behavioral: Weekly Motivational Emails
- Varenicline (Experimental): Varenicline tartrate (Champix®), Pfizer Canada Inc., Kirkland, Quebec. Dispense for 12 weeks. One tablet (0.5mg) once daily for first three days, then one tablet (0.5 mg) twice daily for next four days, then 1 mg (one 1mg tablet or two 0.5mg tablets) twice daily for the remainder of 12 weeks.
  Interventions: Drug: Varenicline; Behavioral: Weekly Motivational Emails

INTERVENTIONS:
Drug: Bupropion
  Arms: Bupropion
Drug: Varenicline
  Arms: Varenicline
Behavioral: Weekly Motivational Emails — The e-mails will include tips on several things other than the medications that participants can do to help them quit smoking. The contents of the emails will vary from week to week. The e-mails will provide tips on ways to create an atmosphere that promotes quitting and staying abstinence. They will also include recommendations on how to address issues with withdrawal symptoms and cravings. In addition, they will provide positive motivational messages by stating facts on benefits of quitting smoking.

SUMMARY:
Clinically proven medications such as nicotine replacement therapy, bupropion and varenicline are available to help smokers quit but there are not widely used. The primary objective of this study is to evaluate the real-world long-term effectiveness of of bupropion and varenicline treatment in a community sample of smokers interested in quitting. The investigators hypothesize that varenicline treatment will result in higher quit rates at end of treatment and at one year after treatment compared to bupropion. Smoking status will be biochemically confirmed at various time points using salivary cotinine measures. Furthermore, since 50% of the variation in quit success is genetically determined, and the effectiveness of different cessation medication may differ considerably in sub-groups of smokers carrying certain genetic variants, the investigators will collect saliva samples from consenting participants to evaluate the moderating effect of genetics on treatment response.

DETAILED DESCRIPTION:
Only a fraction of smokers receive information about effective prescription-only smoking pharmacotherapies, bupropion and varenicline. Moreover, studies have demonstrated variable smoking cessation treatment outcomes correlate with individuals' genotypes and phenotypes. Mass distribution approaches, bypassing clinics and physicians, have been successful for nicotine replacement therapy. The primary objective of this study is to evaluate the real-world long-term effectiveness of mailed bupropion and varenicline treatment in a sample of interested smokers, utilizing web-based recruitment and follow-up. As part of the Genetics Sub-study, the pharmacogenetics of these smoking cessation medications is investigated. This is an open label study, wherein eligible participants will be randomized to receive bupropion (Zyban®) or varenicline (Champix®) for 12 weeks in conjunction with weekly motivational emails. Participants will spend approximately 20-30 minutes enrolling in the study through the study's website. During this time, they will read the consent form, answer the eligibility questions and complete the baseline questionnaire. Eligible participants are then asked if they are interested to participate in the Genetics Sub-study. Those who provide separate consent for the genetics component will complete additional questionnaires online (Between Facets and Domains Personality Test) and will be mailed a kit to provide a saliva sample. After successful completion of baseline questionnaire through the study website, eligible participants will be emailed a Letter to Doctor and a Standard Script to take to their doctor. Then, they will attend an appointment with their physician to discuss with their doctor whether the medication they have been assigned to is appropriate for them to use as smoking cessation aid. It is possible that the participant and his/her doctor will decide not to pursue smoking cessation using the assigned medication. These participants will still receive the weekly motivational emails and will be followed up at all time points, but they will not be included in the main data analysis. If the doctor believes that it is appropriate for the participants to take the assign medication, he/she will need to sign the Standard Script and fax it to the study contract pharmacy. Once the fax is received by the pharmacy, they will call the participants for a brief counseling. Then, they will fill the prescription and mail the medication to you free of charge. All participants will set a quit date of their choosing, but will start the medication 7 days prior to their target quit date. Data related to the outcome measures and adverse events will be collected at 4, 8 and 12, 26 and 52 weeks after the start of treatment in order to assess and compare both point prevalent and continuous abstinence effects of the two treatment interventions. Smoking status will be biochemically confirmed at baseline and at 26th and 52nd weeks following start of treatment using salivary cotinine measures. Medication compliance is assessed by self-report measures as part of the follow-up questionnaire. Compliance is also biochemically confirmed at 4 weeks following start of treatment.

ELIGIBILITY:
Inclusion Criteria:

* At least 19 years of age
* Smoking at least 10 cigarettes per day
* Smoked daily for at least the past year
* Have an intention of quit smoking in the next 30 days.

Exclusion Criteria:

* History of psychotic disorder or eating disorder
* Brain injury
* Seizure disorder
* Pregnancy, lactation, or at risk of becoming pregnant
* Allergy or sensitivity to bupropion or varenicline
* Taking monoamine oxidase inhibitors (anti-depressants), thioridazine or Wellbutrin or other medication containing bupropion hydrochloride.

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 968 (Actual)
Dates: Start 2014-05-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Change in smoking status over time | At 12, 26, and 52 weeks following start of treatment
  Related to effectiveness of smoking cessation intervention, The 7-day point prevalence abstinent rate is defined as not having smoked, even a puff, over the previous seven days.

SECONDARY OUTCOMES:
Pre-post Decisional Balance Scores | upon first patient enrolled and 1 month following last patient enrolled
  Related to physician practice changes after being approached by their patients about smoking cessation medications and being informed about the study.
Continuous Abstinence | 12, 26 and 52 weeks after start of treatment
  A measure of long-term smoking cessation and time to relapse.

OTHER OUTCOMES:
Genetic Polymorphisms | About 5 weeks following participants' enrollment
  Polymorphisms in genes involved in treatment medication and nicotine's metabolism and receptors, as well as genetic variations involved in dopamine neurotransmitter pathway are investigated. DNA analysis is performed using mailed-in saliva samples.
Personality Traits | At baseline
  The ten aspects of personality traits (2 aspects for each big five domains of personality), as described by BFAS (Big Five Aspect Scales), are measured.

CONTACTS AND LOCATIONS:
Overall Officials: Laurie Zawertailo, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Nicotine Dependence Clinic, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Zhang H, Mansoursadeghi-Gilan T, Hussain S, Veldhuizen S, Le Foll B, Selby P, Zawertailo L. Evaluating the effectiveness of bupropion and varenicline for smoking cessation using an internet-based delivery system: A pragmatic randomized controlled trial (MATCH study). Drug Alcohol Depend. 2022 Mar 1;232:109312. doi: 10.1016/j.drugalcdep.2022.109312. Epub 2022 Feb 9. PMID 35151504
- [Derived] Zawertailo L, Mansoursadeghi-Gilan T, Zhang H, Hussain S, Le Foll B, Selby P. Varenicline and Bupropion for Long-Term Smoking Cessation (the MATCH Study): Protocol for a Real-World, Pragmatic, Randomized Controlled Trial. JMIR Res Protoc. 2018 Oct 18;7(10):e10826. doi: 10.2196/10826. PMID 30341043
- See also: Link Text: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addiction teaching hospital. It is fully affiliated with the University of Toronto, and is a PAHO/WHO Collaborating Centre — http://www.camh.net/research